CLINICAL TRIAL: NCT05959954
Title: Quantitative Sensory Testing to Predict Progression to Nociplastic Pain in Carpal Tunnel Syndrome: A Prospective Cohort Study
Brief Title: Predicting Nociplastic Pain in Carpal Tunnel Syndrome Through Quantitative Sensory Testing
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Other Study IDs: CTS-QST-2023
Record Dates: First submitted 2023-07-18; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Carpal Tunnel Syndrome (CTS) Patients: Adults with clinical and electrodiagnostic evidence of carpal tunnel syndrome.
  Interventions: Diagnostic Test: Quantitative Sensory Testing (QST)

INTERVENTIONS:
Diagnostic Test: Quantitative Sensory Testing (QST) — Quantitative Sensory Testing (QST) is a non-invasive diagnostic method used to assess sensory dysfunction. The test evaluates individual thresholds and pain responses to different types of mechanical, thermal, and electrical stimuli. For this study, QST will be used to gather baseline sensory data for patients with carpal tunnel syndrome. This information will then be used to predict the progression to nociplastic pain over a one-year follow-up period.

SUMMARY:
This study aims to investigate the predictive value of quantitative sensory testing (QST) in identifying patients with carpal tunnel syndrome (CTS) who are at risk of developing nociplastic pain.

DETAILED DESCRIPTION:
The study will recruit 120 adults diagnosed with CTS and conduct baseline QST measures. The progression to nociplastic pain will be assessed over a one-year follow-up period to determine the predictive value of QST measures.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18-60
* Clinical diagnosis of CTS based on presence of parasthesias and/or pain in median nerve distribution, positive Phalen's test and/or Tinel's sign, and nocturnal symptoms
* Electrodiagnostic evidence of median neuropathy at the wrist:

  1. Prolonged median motor distal latency >4.2 ms
  2. Prolonged median sensory latency >3.4 ms
* Symptom duration between 6 months and 2 years (to exclude very early or very late stages)
* Pain severity of ≥5 on 0-10 numerical rating scale
* No evidence of thenar muscle atrophy on physical exam
* No prior surgery or fracture of the affected wrist
* No evidence of comorbid diabetes mellitus, cervical radiculopathy, polyneuropathy, or other neuromuscular disorders

Exclusion Criteria:

* Diabetes mellitus, as a common cause of polyneuropathy, which can confound QST measures.
* Cervical radiculopathy or other upper limb neuropathies, which can cause overlapping sensory symptoms and signs.
* History of wrist fracture or surgery, which may cause structural abnormalities affecting nerve function.
* Pregnancy, due to physiological changes that can affect nerve function.
* Patients with severe thenar muscle atrophy, indicating long-standing severe median neuropathy.
* Patients unable to provide informed consent or comply with study procedures.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults with clinical and electrodiagnostic evidence of carpal tunnel syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-07-21 (Estimated); Primary Completion 2024-07-21 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Progression to Nociplastic Pain | 1 year from the start of the study
  Development of nociplastic pain in patients with carpal tunnel syndrome, as identified by a Kosek, by clinical criteria suggest by E., Clauw, D., Nijs, J., Baron, R., Gilron, I., Harris, R. E., ... & Sterling, M. (2021). Chronic nociplastic pain affecting the musculoskeletal system: clinical criteria and grading system. Pain, 162(11), 2629-2634.

SECONDARY OUTCOMES:
Change in Quantitative Sensory Testing (QST) Measures | Changes in QST at baseline and 1 year
  A significant change in QST measures could indicate the progression of sensory abnormalities in the participants. QST measures include thermal detection and pain thresholds, mechanical detection and pain thresholds, and vibration detection thresholds. Each of these thresholds is measured using specific testing equipment and protocols, and the exact scoring can vary based on the specific equipment and protocol used. In general, lower thresholds (i.e., the patient detects the stimulus at lower intensities) may indicate heightened sensitivity or hyperalgesia, while higher thresholds may indicate reduced sensitivity or hypoesthesia. Changes in these thresholds over time can indicate a worsening of sensory dysfunction.

OTHER OUTCOMES:
Change in Hand Function | Change in hand function measures at baseline and 1 year.
  Hand function can be measured using tools like the Boston Carpal Tunnel Questionnaire, which includes two scales: the Symptom Severity Scale and the Functional Status Scale. The Symptom Severity Scale measures the severity and frequency of symptoms, while the Functional Status Scale measures the impact of these symptoms on daily activities. Each item on these scales is rated on a scale of 1 (no symptoms or difficulty) to 5 (most severe symptoms or difficulty). Higher scores on the Symptom Severity Scale and lower scores on the Functional Status Scale indicate worse hand function. An increase in the Symptom Severity Scale score or a decrease in the Functional Status Scale score over time would indicate a worsening of hand function.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Chair — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No